CLINICAL TRIAL: NCT01121068
Title: Monthly Follow up of Interferon Gamma Releasing Assay Among Health-care Workers Treating TB Patients
Brief Title: Monthly Follow up of Interferon Gamma Releasing Assay (IGRA) Among Health-care Workers Treating Tuberculosis (TB) Patients
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Joon Yim, Professor, Seoul National University Hospital
Other Study IDs: monthly IGRA
Record Dates: First submitted 2010-05-09; First posted 2010-05-12 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Tuberculosis
Keywords: IGRA; variability; Long-term variability of IGRA
MeSH Terms: conditions — Tuberculosis | interventions — Cordocentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Health care workers
  Interventions: Other: Blood samplings

INTERVENTIONS:
Other: Blood samplings — About 3.5ml of blood will be drawn from the participants monthly.

SUMMARY:
Interferon gamma releasing assay(IGRA) is useful to diagnose latent tuberculosis. However,IGRA responses could show within-subject variability. We wanted to determine long-term IGRA variability in health-care workers who continuously expose to tuberculosis patients.

DETAILED DESCRIPTION:
IGRA will be performed monthly in health-care workers with continuous exposure to tuberculosis patients for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Health care workers who are continuously exposed to TB patients Age > 20 years

Exclusion Criteria:

* Pregnant Active TB Use of immunosuppressants

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care workers who are continuously exposed to TB patients
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Results of interferon-gamma releasing assay | monthly for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, Study Chair — Division of Pulmonology and Critical Care Medicine, Department of Internal Medicine and Lung Institute of Medical Research Center, Seoul National University College of Medicine
Locations (1):
- Division of Pulmonology and Critical Care Medicine, Department of Internal Medicine and Lung Institute of Medical Research Center, Seoul National University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Park JS, Lee JS, Kim MY, Lee CH, Yoon HI, Lee SM, Yoo CG, Kim YW, Han SK, Yim JJ. Monthly follow-ups of interferon-gamma release assays among health-care workers in contact with patients with TB. Chest. 2012 Dec;142(6):1461-1468. doi: 10.1378/chest.11-3299. PMID 22556318